CLINICAL TRIAL: NCT01511549
Title: A Randomized, Double-blind, Placebo-controlled Ascending Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SAR113945 (IKK Inhibitor) Following Intra-articular Administration in Japanese Patients With Knee Osteoarthritis
Brief Title: Safety, Tolerability and Pharmacokinetics of SAR113945 in Japanese Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDU11333; U1111-1121-4499 (Other: UTN)
Record Dates: First submitted 2012-01-06; First posted 2012-01-18 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 (Experimental): SAR113945 low dose
  Interventions: Drug: SAR113945
- Dose 2 (Experimental): SAR113945 medium dose
  Interventions: Drug: SAR113945
- Dose 3 (Experimental): SAR113945 high dose
  Interventions: Drug: SAR113945
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Pharmaceutical form:injection
  Route of administration: intra-articular
  Arms: Placebo
Drug: SAR113945 — Pharmaceutical form:injection
  Route of administration: intra-articular
  Arms: Dose 1; Dose 2; Dose 3

SUMMARY:
Primary Objective:

To assess the safety and tolerability of SAR113945 in Japanese patients with knee osteoarthritis after ascending single intra-articular doses

Secondary Objective:

To assess the pharmacokinetics of SAR113945 in Japanese patients with knee osteoarthritis after ascending single intra-articular doses

DETAILED DESCRIPTION:
Following the single dose of study medication, the study period for each patient will be 168 days.

ELIGIBILITY:
Inclusion criteria:

* Japanese male or female patients, aged 40 years or older, with knee osteoarthritis
* Diagnosis of primary knee osteoarthritis, based upon the following:

  * X-ray or magnetic response imaging (MRI) evidence within the last 6 months for joint space narrowing and osteophyte formation
  * Patients will be Kellegen and Lawrence classification II or III, and total Western Ontario McMaster (WOMAC) score below or equal to 72
  * Patients fulfilling the American College of Rheumatology Clinical and Radiographic criteria for Osteoarthritis

Exclusion criteria:

* Women of child bearing potential
* Secondary osteoarthritis: e.g., autoimmune disease, joint dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos syndrome, Gaucher's disease, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, calcium pyrophosphate disposition disease, or neuropathic arthropathy
* Presence of local skin abnormality at the affected knee joint
* Any patient who received intra-articular injection within 3 months prior to administration

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with safety assessments (adverse events, vital signs, 12 lead ECGs and laboratory tests) | up to 24 weeks
Examination of skin/soft tissue of injected knee, and knee joint | up to 24 weeks
  Examination of skin/soft tissue of injected knee: Any reaction is classified as erythema, edema, pain, hematoma and graded none, mild, moderate or severe.
  Examination of knee joint of injected knee: Any reaction is classified as effusion/worsening of effusion, warmth and pain.

SECONDARY OUTCOMES:
Pharmacokinetic parameter (AUC) | 21 time points up to 24 weeks
Pharmacokinetic parameter (Cmax) | 21 time points up to 24 weeks
Pharmacokinetic parameter (tmax) | 21 time points up to 24 weeks
Pharmacokinetic parameter (t1/2) | 21 time points up to 24 weeks
Pharmacodynamic parameter (WOMAC index) | up to 24 weeks
Pharmacodynamic parameter (biomarkers relating to osteoarthritis) | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 392001, Osaka, Japan